CLINICAL TRIAL: NCT04057079
Title: Anugel vs Gelatine Sponge Clinical Trial
Brief Title: Comparing Anugel With Gelatine Sponges for Pain Management After Hemoroidectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Deep Life Medical Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Anugel20170420
Record Dates: First submitted 2019-05-01; First posted 2019-08-15 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Pain, Postoperative
Keywords: Hemoroidectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Research staff used a computer-based tool to allocate the ligasure haemorrhoidectomy patients randomly to either Group 1 (n=56) who received standard anal gelatine sponge (SpongostanTM) or Group 2 (n-54) to a layered hydrogel sponge (AnugelTM) following surgery. Encryption concealed the allocation until the patient's details had been logged.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anugel (Experimental): In this arm, after the surgery a hydrogel impregnated sponge will be placed in the rectum.
  The patient is evaluated after the operation and the following day when the sponge is removed.
  A hydrogel impregnated foam pad is applied on the surface of the wound the following 5 days.
  The patient is evaluated on post op, on day 1 (usually before discharge) and day 5
  The pain of the patients are evaluated according to the VAS scale and the use of analgesics and opioids is monitored.
  Interventions: Combination Product: Anugel, Hydrogel sponge
- Sponge (Active Comparator): Currently used treatment method i.e. insertion of gelatine sponge in to the rectum post operation.
  The patient is evaluated on post op, on day 1 (usually before discharge) and day 5
  The pain of the patients are evaluated according to the VAS scale and the use of analgesics and opioids is monitored.
  Interventions: Combination Product: Gelatine Sponge

INTERVENTIONS:
Combination Product: Anugel, Hydrogel sponge — A calibrated sponge impregnated with hydrogel is inserted to the rectum post hemoroidectomy.
  Arms: Anugel
Combination Product: Gelatine Sponge — A gelatine sponge is inserted in to the rectum pos hemoroidectomy.
  Arms: Sponge

SUMMARY:
Post-operational pain is the most common problem relating to haemorrhoidectomy. This study aims to evaluate the postoperative effects of Anugel a hydrogel impregnated multi component sponge vs gelatine sponge comparatively.

DETAILED DESCRIPTION:
The patients were placed in the lithotomy position. Haemorrhoids (piles) were later located through exploration. The piles were dissected using ligasure. After completing the dissection, bleeding was controlled and either Anugel or the gelatine sponge (SpongostanTM) is inserted in to the rectum as determined by patient allocation.

The patients were monitored post operation and 5 days following the surgery. Pain was measured using the VAS scale and use of pain medication was monitored.

ELIGIBILITY:
Inclusion Criteria:

* Haemorrhoid (grade 3-4)

Exclusion Criteria:

* Repeating cases, additional (non haemorrhoid related) complications

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-04-04 (Actual); Primary Completion 2018-07-09 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Pain Reduction | 5 days
  Amount of pain patients feel post operation. Post surgery and on days 1 and 5 the pain felt by the patient will be measured according to the VAS scale, either in hospital or during hospital visit.

SECONDARY OUTCOMES:
Use of analgesics | 5 days
  The frequency and dose of analgesics for pain management is monitored post operation, on day 1 and day 5

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Sisli Hospital, Istanbul, Sisli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided